CLINICAL TRIAL: NCT02603003
Title: A Study on the"Fuzheng"Therapy Promoted Immune Reconstitution to Improve the Survival of Early-stage Lung Cancer After Surgical Operation
Brief Title: the"Fuzheng" Therapy of TCM to Improve the Survival Quality of Early-stage NSCLC by Intervening the CTCs
Acronym: CTC-TCM-FZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, jianhuitian, Clinical Professor, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Longhua Hospital; TJH20151021 (Registry Identifier: TIAN Jianhui); LB20151106 (Registry Identifier: Robin)
Record Dates: First submitted 2015-10-21; First posted 2015-11-11 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Non-small Cell Lung Cancer(NSCLC)
Keywords: Circulating tumor cells(CTCs); Traditional Chinese Medicine(TCM); Myeloid-derived suppressor cells(MDSCs)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating | interventions — jinfukang; Cisplatin; Vinorelbine; Pemetrexed; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cisplatin (Placebo Comparator): Cisplatin
  Interventions: Drug: Cisplatin
- Pemetrexed (Placebo Comparator): Pemetrexed
  Interventions: Drug: Pemetrexed
- Jinfukang (Experimental): Jinfukang
  Interventions: Drug: JinFuKang; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: JinFuKang — po.tid.30ml
  Other Names: Jin Fukang oral liquid
  Arms: Jinfukang
Drug: Cisplatin — According to the individual patient's condition
  Other Names: Navelbine
  Arms: Cisplatin; Jinfukang
Drug: Pemetrexed — According to the individual patient's condition
  Other Names: Pemetrexeddisodium for Injection
  Arms: Jinfukang; Pemetrexed

SUMMARY:
Metastasis is the leading cause of death in patients with lung cancer, and circulating tumor cells(CTCs) play a key role in the process of distant metastasis. The investigators' study will elaborate the clinical significance of CTCs intervented by Traditional Chinese Medicine(TCM) in lung cancer from the diagnosis and clinical staging,metastasis and recurrence, individual treatment and prognosis and so on, in order to provide a new direction for the treatment of lung cancer.

DETAILED DESCRIPTION:
Metastasis is the leading cause of death in patients with lung cancer, and circulating tumor cells play a key role in the process of distant metastasis.In recent years, research results have shown that CTCs may become a emerging marker and new target in the treatment of lung cancer. The investigators' study will elaborate the clinical significance of CTCs intervented by TCM in lung cancer from the diagnosis and clinical staging,metastasis and recurrence, individual treatment and prognosis and so on, in order to provide a new direction for the treatment of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Complete resection was accepted in IIa ~ Ⅲa stage, and the pathological changes could confirmed as non small cell lung cancer patients;
2. Patients receiving chemotherapy for the first time in 6 weeks after surgery;
3. Age from 18 Years to 70 Years;
4. The liver and renal function were normal,and no other disease.
5. Patients compliance is good ang can understand the situation of this study and signed informed consent

Exclusion Criteria:

1. Patients without clear pathological diagnosis;
2. The expected survival period is morn than 6 months;
3. Patients with serious diseases such as heart, liver, kidney and hematopoietic system;
4. Patients with pregnancy or lactation;
5. Persons with a history of less control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2015-06; Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | The progression disease is assessed based on CT or PET-CT every six months from date of randomization and the endpoints is the date of first documented progression or date of death due to lung cancer,assessed up to Two years.
  It is decided by a doctor via the clinical examinations

SECONDARY OUTCOMES:
Circulating Tumor Cell | 24months
  It is decided by a doctor via the clinical examinations
Overall survival | Two years
  It is decided by a doctor via the clinical examinations